CLINICAL TRIAL: NCT06173414
Title: Adaptive Optics ScanningLaser Ophthalmoscope Safety and Efficacy Clinical Trial
Status: Completed | Type: Observational
Sponsor: Robotrak Technologies Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: RT-MONA-2023-01
Record Dates: First submitted 2023-11-22; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Retinal Disease; Healthy
Keywords: healthy patients; eye disease
MeSH Terms: conditions — Retinal Diseases; Eye Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention measures — No intervention measures

SUMMARY:
This prospective, multicenter, single-group, target-value clinical trial was designed to evaluate the efficacy and safety of an Adaptive Optics ScanningLaser Ophthalmoscope(AOSLO) for ophthalmic examination.

DETAILED DESCRIPTION:
objective: This study aims to collect AOSLO retinal images from human population to assess the imaging quality and quantitative measurement consistency of AOSLO devices manufactured by Robotrak and also monitor any possible side effects.

study population: randomly invited 194 volunteers who meets inclusion criteria

design: the study is an observational protocol that participants will be imaged with Robotrak AOSLO systems to get cellular level images of photoreceptors and blood vessels in foveal area. Automatics analysis of cell/blood vessel morphology parameters will be calculated for consistency evaluation. In general, participants will undergo a complete ophthalmic examination including assessments of visual acuity, intraocular pressure, slit lamp examination, ocular biometry, OCT, fundus imaging, multi-focal ERG and OCT scan to assess potential side effects of AOSLO imaging.

outcome measures: the primary efficacy outcome measure of this study are multi expert grading of the image quality collected.

the secondary efficacy outcome measure are quantitative assessment of the morphological parameters generated from the captured images and device operator ratings.

the safety measures are side effect signs from ophthalmic examinations before&after AOSLO imaging

ELIGIBILITY:
Inclusion criteria：

1. Age range from 18 to 65 years old (including 18 and 65 years old), regardless of gender;
2. Can fully cooperate with instructions to complete the inspection
3. The subject (or their designated agent) voluntarily participates and signs an informed consent form. Note: At least 63 subjects with no obvious eye abnormalities were enrolled (determined by the researcher through ophthalmic examination)

exclusion criteria：

1. Patients with high intraocular pressure (>21mmHg) or other reasons who cannot undergo mydriasis;
2. For those with a spherical lens degree exceeding 5D or a cylindrical lens degree exceeding ± 2D,
3. those with ptosis or other conditions that cannot fully expose the pupil area
4. Aphthalmic or intraocular lens eyes
5. Those who have received photodynamic therapy within 48 hours;
6. Individuals with a history of photosensitivity or taking medication that may cause photosensitive side effects 7）Those who have obvious skin lesions on the lower jaw or forehead and are unable to contact the lower jaw or forehead support

8) Individuals with epidemic keratoconjunctivitis or in the active phase of other infectious diseases 9) Those whose refractive medium is turbid and unable to obtain satisfactory images; 10) Poor fixation or inability to cooperate with the examination due to other reasons; 11) Pregnant or lactating women;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: randomly invited volunteers from primary eyecare outpatient patients or accompanying family members who meet the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-11-16 (Actual)

PRIMARY OUTCOMES:
Image quality excellence rate | through study completion, an average of half year
  Divide the collected images into 25 small squares based on a 5X5 square grid; Divide each small square into "clear" and "under clear" based on whether the mosaic structure of photosensitive cells is clear and visible. Divide the entire 2.4 ° X2.4 'image into three levels: "excellent", "good", and "poor" based on the proportion of small squares evaluated as "clear" among the 25 squares in each image: "excellent" is defined as the proportion of "clear" small squares ≥ 80%; The definition of "good" image quality is that the proportion of "clear" small squares is>60% but<80%; The definition of "poor" image quality is that the proportion of "clear" small squares is less than 60%; Calculate the proportion of images with "excellent" and "good" imaging quality to all images.

SECONDARY OUTCOMES:
Repeatability of cell analysis function | through study completion, an average of half year
  The Adaptive Optics ScanningLaser Ophthalmoscope by Robotrak Technologies Co., Ltd. has image post-processing function, which can analyze single cell images, generate photoreceptor cell density, photoreceptor cell spacing, photoreceptor cell regularity, and photoreceptor cell dispersion. The operator collected images of the photoreceptor cell layer from three positions in the subject's retina (8.8 ° above the fovea of the macula and 8.8 ° below the fovea of the macula), with 5 independent images collected from each position. Repeatability evaluation using ICC intra group correlation coefficients after removing the highest and lowest values.
Repeatability of vascular blood flow analysis function | through study completion, an average of half year
  The Adaptive Optics ScanningLaser Ophthalmoscope by Robotrak Technologies Co., Ltd. can obtain quantitative blood flow indicators such as vascular wall thickness, vascular diameter, lumen diameter, wall/lumen ratio, vascular wall cross-sectional area, and blood flow velocity. The operator collected 5 independent images of the subject's retina at the same position and vascular level, and recorded the above information generated by the machine. After removing the highest and lowest values, the ICC intra group correlation coefficient was used to evaluate repeatability.
Satisfaction rate of device performance and operational evaluation | through study completion, an average of half year
  The operator evaluates the performance and operation of the device on a scale based on the usage situation after the inspection is completed.
Satisfaction rate of clinical function and applicability evaluation of devices | through study completion, an average of half year
  The operator evaluates the clinical function and applicability of the adaptive optical fundus imaging system for fundus examination using a scale based on usage.
Adverse event occurrence rate | through study completion, an average of half year
  The incidence of adverse events, including but not limited to the following possible adverse events:
  Eye surface damage: During multifocal electroretinogram examination, corneal electrodes need to be worn on the cornea, which may cause eye surface damage. If corneal injury or severe conjunctival congestion occurs, topical eye drops can be used to combat infection and promote corneal epithelial repair.
  Eye fatigue: During the examination process, subjects may experience eye fatigue due to measuring the brightness of the light source. Generally, it can improve after a brief rest Infection: Due to insufficient cleaning and disinfection of the collar and forehead pads under the device, repeated use may cause cross infection of the subject's skin. Once an infection is detected, symptomatic treatment is sufficient.

CONTACTS AND LOCATIONS:
Overall Officials: Qian Liu, O.D., Principal Investigator — Henan Provincial Eye Hospital
Locations (1):
- Robotrak Technologies Co., Ltd., Nanjing, China

IPD SHARING:
Plan to Share IPD: No
Not yet decided